CLINICAL TRIAL: NCT06369714
Title: Neurofeedback-Based Digital Therapeutics for the Diagnosis and Treatment of Attention Deficit Hyperactivity Disorder (ADHD) in Children.
Brief Title: Neurofeedback-Based Digital Therapeutics for the Diagnosis and Treatment of ADHD in Children.
Acronym: ADHD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lei Lei, MD (Other)
Responsible Party: Sponsor-Investigator, Lei Lei, MD, Associate Chief Physician, Principal Investigator, Changhai Hospital
Organization: Changhai Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHEC2023-296
Record Dates: First submitted 2024-04-02; First posted 2024-04-17 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Attention Deficit Disorder With Hyperactivity; Executive Function Disorder
Keywords: Digital Therapeutics; Neurofeedback; Attention Deficit Disorders with Hyperactivity; Children; Executive function disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Medication group (Active Comparator): The medication group will take Methylphenidate Hydrochloride Extended-Release Tablets with a fixed dose for eight weeks.
  Interventions: Drug: Concerta
- Digital therapeutics group (Experimental): The digital therapeutics group will complete 30 training sessions within 8 weeks.
  Interventions: Device: Digital therapeutics
- Combination group (Experimental): The combination group will take Methylphenidate Hydrochloride Extended-Release Tablets while undergoing digital therapeutics.
  Interventions: Drug: Concerta; Device: Digital therapeutics

INTERVENTIONS:
Drug: Concerta — Methylphenidate Hydrochloride Extended-Release Tablets with the following specifications: 18mg dosage, oral administration, once a day for a duration of 8 weeks.
  Other Names: Methylphenidate Hydrochloride Extended-Release Tablets
  Arms: Combination group; Medication group
Device: Digital therapeutics — 30 sessions of digital therapeutics, each lasting 30 minutes, will be conducted with a frequency of once every 1-2 days over an 8-week period.
  Arms: Combination group; Digital therapeutics group

SUMMARY:
A multi-center, randomized controlled trial is being conducted to investigate the efficacy of a novel digital therapeutics (DTx) program that utilizes a cross-training approach between neurofeedback training and executive function training for pediatric patients (aged 6-12) diagnosed with ADHD. This gamified interactive program is designed to improve attention deficits and executive function impairments in pediatric patients with ADHD. It is delivered through an engaging iPad game in a home-based treatment format. Patients will be randomly assigned to one of three groups: medication alone, digital therapeutics alone, or a combination of both interventions. Subjects will undergo 30 treatment sessions over the 8-week period, with each session lasting 30 minutes. Investigators will reassess symptoms of ADHD, executive functions, and objective measures of attention at the end of the treatment. Additionally, questionnaires will be distributed to parents to gather their insights and feedback on the treatment approach. This innovative digital therapeutics approach is expected to improve ADHD symptoms individually and enhance therapeutic outcomes when used alongside conventional drug treatment regimens.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria established by the 5th edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) for ADHD.
* Digital Cancellation Test total score<50 points.
* Raven's Standard Progressive Matrices score≥85.
* 6 years ≤ Age<12 years.
* No interventions for ADHD received within 4 weeks.
* No color blindness.

Exclusion Criteria:

* Patients with organic mental disorders, schizophrenia, bipolar disorder, depressive disorders, and other psychiatric conditions.
* Patients with comorbid autism spectrum disorder, Tourette's syndrome, and other neurodevelopmental disorders.
* Patients with comorbid conduct disorders.
* Patients with severe traumatic brain injury or neurological disorders.
* Patients with a history of severe somatic diseases.
* Patients with a history of substance or drug dependency.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 210 (Estimated)
Dates: Start 2023-02-24 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Swanson, Nolan, and Pelham IV Rating Scale | Baseline to End of Treatment (Week 8) and to Follow-up (Week 20, Week 32)
  The Swanson, Nolan, and Pelham IV Rating Scales (SNAP-IV) will be completed by parents to assess the severity of ADHD symptoms. The values range from 0 to 3, with lower scores indicating a better outcome.

SECONDARY OUTCOMES:
Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition criteria for ADHD | Baseline to End of Treatment (Week 8) and to Follow-up (Week 20, Week 32)
  The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for ADHD will be used to assess the number of core symptoms. There are a total of 18 core symptoms, with fewer symptoms indicating a better outcome.
Questionnaire-Children with Difficulties | Baseline to End of Treatment (Week 8) and to Follow-up (Week 20, Week 32)
  The Questionnaire-Children with Difficulties (QCD) will be completed by parents to assess the social abilities of participants. The total questionnaire score is 57, and a score below 30 suggests impaired functioning.
Behavior Rating Inventory of Executive Function | Baseline to End of Treatment (Week 8) and to Follow-up (Week 20, Week 32)
  The Behavior Rating Inventory of Executive Function (BRIEF) will be completed by parents to assess changes in executive function. The normal standards for scores vary by age, with lower scores indicating a better outcome.
Continuous Performance Test | Baseline to End of Treatment (Week 8) and to Follow-up (Week 20, Week 32)
  A newly designed Continuous Performance Test (CPT) will be administered to participants by investigators, with higher accuracy rates indicating a better outcome.
Digital Cancellation Test | Baseline to End of Treatment (Week 8) and to Follow-up (Week 20, Week 32)
  The Digit Cancellation Test (DCT) will be administered to participants by investigators, with higher scores indicating a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Lei, MD, Principal Investigator — Department of Pediatric, Changhai Hospital, Naval Medical University
Locations (2):
- China (2):
  - Changzheng Hospital, Naval Medical University, Shanghai, Shanghai Municipality
  - Changhai Hospital, Naval Medical University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No